CLINICAL TRIAL: NCT02620631
Title: Prospective, Randomized, Double-blinded, Placebo-controlled Study to Examine Pain Relief and the Need for Supplementary Analgesics With Intra-thecal Morphine Sulfate (0.2 mg) in Patients Undergoing Total Knee Arthroplasty (TKA)
Brief Title: Study to Examine Pain Relief With Supplemental Intrathecal Morphine in TKA Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Syed Azim, Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 200362
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Acute Pain
Keywords: Morphine; TKA; Pain; TKR; Arthroplasty
MeSH Terms: conditions — Acute Pain; Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects receive intrathecal injection of saline at time of spinal anesthesia
  Interventions: Drug: Placebo
- Morphine (Experimental): Subjects receive intrathecal injection of morphine sulfate 0.2mg at time of spinal anesthesia
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Subjects receive intrathecal morphine pre-operatively to determine its level of efficacy in acute pain control post-operatively when used in conjunction with post-operative PCA morphine
  Other Names: Preservative-free morphine sulfate
  Arms: Morphine
Drug: Placebo — Subjects receive intrathecal, preservative-free normal saline pre-operatively in conjunction with post-operative PCA morphine
  Other Names: Preservative-free normal saline
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blinded, placebo-controlled study designed to examine pain relief following intrathecal morphine sulfate (0.2mg) in patients undergoing total knee arthroplasty (TKA) under spinal anesthesia in addition to a femoral nerve catheter. The protocol consists of two parts: (1) a prospective patient recruitment study and (2) a retrospective assay for endocannabinoids on previously collected specimens.

DETAILED DESCRIPTION:
This is a prospective, case-controlled randomized, double-blinded, placebo-controlled study expected to enroll up to 100 patients scheduled to undergo unilateral total knee arthroplasty (TKA) under regional anesthesia (defined as intrathecal spinal + femoral nerve blockade + femoral nerve catheter for post-operative analgesia) at Stony Brook Hospital. The patients were randomized to receive either IT morphine 0.2 mg (Group 1) or placebo (Group 2) in combination with their standard-of-care spinal anesthesia. Post-operatively, the patients were given an intravenous patient-controlled analgesic opioid for breakthrough pain.

Only the pharmacist preparing the drug/placebo has knowledge of how each subject was randomized. Study staff completed multiple questionnaires regarding subjects' pain scores and patient disability from pain to assess changes between different study periods (ie. pre-operative, post-operative and follow up). Biological samples were also taken from each subject to measure and analyze differences and changes in endocannabinoid levels.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral TKA under regional anesthesia
* ASA Class 1, 2 or 3
* Able to give informed consent
* Able to understand English

Exclusion Criteria:

* Medical condition(s) that prevents use of regional anesthesia (e.g. infection at site of injection, coagulopathy, severe hypovolemia, severe aortic or mitral stenosis, increased intracranial pressure, severe spinal deformity, spinal cord hardware or stimulator implanted)
* Allergy to morphine
* Morbid obesity (BMI > 45)
* Respiratory compromise (difficult airway, severe emphysema or COPD)
* Obstructive sleep apnea (only if diagnosed in a sleep disorders clinic and CPAP was prescribed)
* Chronic pain with opioid usage over 100 mg morphine-equivalents po/day
* History of abuse of opioids or other drugs of abuse
* Scheduled for bilateral TKA
* Revision of knee arthroplasty
* Any medical condition that would affect the patient's ability to metabolize or excrete the study drugs (e.g. chronic kidney failure with patient on dialysis) or other medical condition that in the investigator's opinion would render the patient unsuitable for this research study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Acute pain at rest | 0-24 hours
  Numerical rating scale pain scores were collected every 4 hours

SECONDARY OUTCOMES:
Total opioids dispensed | 0-24 hours
  Total dosage of opioids (in morphine equivalent doses) measured over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Syed Azim, MD, Principal Investigator — Stony Brook Medicine, Department of Anesthesia
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

REFERENCES:
- [Derived] Kaczocha M, Azim S, Nicholson J, Rebecchi MJ, Lu Y, Feng T, Romeiser JL, Reinsel R, Rizwan S, Shodhan S, Volkow ND, Benveniste H. Intrathecal morphine administration reduces postoperative pain and peripheral endocannabinoid levels in total knee arthroplasty patients: a randomized clinical trial. BMC Anesthesiol. 2018 Feb 27;18(1):27. doi: 10.1186/s12871-018-0489-5. PMID 29486720